CLINICAL TRIAL: NCT00563667
Title: Effect of Pterygium Excision on IOL Power Calculation: Concurrent Cataract and Pterygium
Brief Title: Effect of Pterygium Excision on Intraocular Lens Power Calculation for Subsequent Cataract Operation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Authority, Hong Kong (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2003.353; HARECCTR0500013
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-07

CONDITIONS: Pterygium; Cataract; Astigmatism
Keywords: Pterygium; Cataract; Astigmatism
MeSH Terms: conditions — Pterygium; Cataract; Astigmatism

INTERVENTIONS:
Procedure: pterygium excision

SUMMARY:
Pterygium is known to induce with-the-rule astigmatism. Excision of pterygium will steepen the cornea and reduce corneal astigmatism. We postulate that the alteration of keratometry reading will indirectly affect the IOL power calculation in cases with concurrent pterygium and cataract. Concurrent pterygium and cataract is common in Hong Kong and other tropical regions. The effect of pterygium excision on intraocular lens power calculation is investigated.

ELIGIBILITY:
Inclusion Criteria:

* All cases with concomitant cataract and primary pterygium, which are indicated for surgery.

Exclusion Criteria:

* Pterygium smaller than 1mm, which is not visually significant.
* Double headed pterygium
* Pterygium obscuring visual axis that preclude keratometry or autorefraction measurements.
* Previous corneal refractive surgery that alter the keratometric power of the cornea.
* Patients with medical problems that preclude staged ocular surgery, e.g. dementia, heart disease, on warfarin.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2003-12; Study Completion 2004-12 (Estimated)

PRIMARY OUTCOMES:
IOL power | 1 and 3 months post pterygium excision
Astigmatism | 1 and 3 months post pterygium excision

CONTACTS AND LOCATIONS:
Overall Officials: Lulu Cheng, Dr, Principal Investigator — Department of DOVS, Prince of Wales Hospital/ The Chinese University of Hong Kong
Locations (3):
- China (3):
  - Alice Ho Miu Ling Nethersole Hospital, Hong Kong
  - Hong Kong Eye Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong